CLINICAL TRIAL: NCT05588921
Title: A Deep Learning-based Indicator to Reveal Biological Age Using Lens Photographs
Brief Title: LensAge to Reveal Biological Age
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Professor, Sun Yat-sen University
Other Study IDs: LA-2022
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Ophthalmology; Lens Opacities; Biological Age
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aging group: Participants with baseline information, medical history of diseases, and lens photographs

SUMMARY:
Assessment of aging is central to health management. Compared to chronological age, biological age can better reflect the aging process and health status; however, an effective indicator of biological age in clinical practice is lacking. Human lens accumulates biological changes during aging and is amenable to a rapid and objective assessment. Therefore, the investigators will develop LensAge as an innovative indicator to reveal biological age based on deep learning using lens photographs.

ELIGIBILITY:
Inclusion Criteria:

* ages from 20 to 100 years
* have anterior segment photographs
* have ophthalmic and physical examination records

Exclusion Criteria:

* have a history of previous eye surgery, eye trauma, or ocular diseases that can cause complicated cataracts
* baseline information missing

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants aged 20 to 90 have anterior segment photographs, baseline information, and medical records.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The difference between LensAge and chronological age | Baseline
  The age estimation models based on a convolutional neural network (CNN) using lens photographs will be used to generate LensAge. LensAge at the individual level will be calculated by averaging the results of all images corresponding to one individual. The difference between LensAge at the individual level and chronological age will be used to unveil an individual's aging process. A difference above 0 indicates an individual with a faster pace of aging than their peers of the same chronological age, while a difference below 0 indicates a slower pace of aging.

SECONDARY OUTCOMES:
Correlation between the LensAge difference and age-related health parameters | Baseline
  Age-corrected LensAge differences will be used to investigate the odds ratios (ORs) with age-related health parameters.
Mean absolute error (MAE) of the DL age estimation model. | Baseline
  Mean absolute error (MAE) in terms of both image level and individual level will be used to evaluate the performance of the DL age estimation model.
Mean error (ME) of the DL age estimation model. | Baseline
  Mean error (ME) in terms of both image level and individual level will be used to evaluate the performance of the DL age estimation model.
R-squared (R2) of the DL age estimation model. | Baseline
  R-squared (R2) in terms of both image level and individual level will be used to evaluate the performance of the DL age estimation model.

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D., Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity, Guangzhou, Guangdong, China